CLINICAL TRIAL: NCT01627223
Title: Comparison Between Lamivudine and Entecavir Treatment in Patients With Spontaneous Severe Acute Exacerbation of Chronic Hepatitis B.
Brief Title: Comparison Between Lamivudine and Entecavir Treatment in Spontaneous Severe Acute Exacerbation
Acronym: NUC115132
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow progress in recruiting study patients
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Sheng-Shun Yang, M.D. Division of Gastroenterology, Departmemt of Internal Medicine, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUC115132
Record Dates: First submitted 2012-06-18; First posted 2012-06-25 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Hepatitis B
Keywords: Spontaneous Severe Acute Exacerbation of Chronic Hepatitis B; Lamivudine (Zeffix®); Entecavir (Baraclude®)
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamivudine 100 mg p.o. q.d. (Experimental): To target 88 evaluable subjects, approximately 98 patients should be recruited into this trial. After enrollment, all eligible subjects will be randomly assigned to one of the antiviral treatments below.
  * Cohort 1: Lamivudine 100 mg p.o. q.d.
  * Cohort 2: Entecavir 0.5 mg p.o. q.d.
  This process will be stratified by prolonged PT, < 4 sec / 4-6 sec / > 6 sec. Both lamivudine and entecavir will be taken once daily and the first dose of observational drug should be administered on Day 1. The observational period of individual subject will be 12 weeks; however, both treatments could be continued after the end of study based on physician's clinical judgment.
  Interventions: Drug: Lamivudine
- Entecavir 0.5 mg p.o. q.d (Experimental): To target 88 evaluable subjects, approximately 98 patients should be recruited into this trial. After enrollment, all eligible subjects will be randomly assigned to one of the antiviral treatments below.
  * Cohort 1: Lamivudine 100 mg p.o. q.d.
  * Cohort 2: Entecavir 0.5 mg p.o. q.d.
  This process will be stratified by prolonged PT, < 4 sec / 4-6 sec / > 6 sec. Both lamivudine and entecavir will be taken once daily and the first dose of observational drug should be administered on Day 1. The observational period of individual subject will be 12 weeks; however, both treatments could be continued after the end of study based on physician's clinical judgment.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Lamivudine — Lamivudine 100 mg p.o. q.d.
  This process will be stratified by prolonged PT, < 4 sec / 4-6 sec / > 6 sec. Both lamivudine and entecavir will be taken once daily and the first dose of observational drug should be administered on Day 1. The observational period of individual subject will be 12 weeks; however, both treatments could be continued after the end of study based on physician's clinical judgment.
  Other Names: Zeffix®
  Arms: Lamivudine 100 mg p.o. q.d.
Drug: Entecavir — •Entecavir 0.5 mg p.o. q.d
  This process will be stratified by prolonged PT, < 4 sec / 4-6 sec / > 6 sec. Both lamivudine and entecavir will be taken once daily and the first dose of observational drug should be administered on Day 1. The observational period of individual subject will be 12 weeks; however, both treatments could be continued after the end of study based on physician's clinical judgment.
  Other Names: Baraclude®
  Arms: Entecavir 0.5 mg p.o. q.d

SUMMARY:
This is a prospective, observational, open-label, 2-arm, parallel, multi-center study. Patients with HBV-associated severe acute exacerbation for whom the treatment with NRTI (such as lamivudine and entecavir) is medically recommended will be screened for eligibility. To target 74 evaluable subjects, approximately 82 patients should be recruited into this trial. After enrollment, all eligible subjects will be randomly assigned to one of the antiviral treatments below.

* Cohort 1: Lamivudine 100 mg p.o. q.d.
* Cohort 2: Entecavir 0.5 mg p.o. q.d. This process will be stratified by prolonged PT, < 4 sec / 4-6 sec / > 6 sec. Both lamivudine and entecavir will be taken once daily and the first dose of observational drug should be administered on Day 1. The observational period of individual subject will be 12 weeks; however, both treatments could be continued after the end of study based on physician's clinical judgment.

The efficacy and safety data will be collected at baseline, 3, 5, 8, 15, 22, 29, 85, and 180 days after initiation of antiviral treatment. All assessments should be conducted based on routine practice of each hospital. Only the analysis of HBV DNA and anti-HDV will be performed in the central lab. For patients who are willing to provide the residual samples of HBV DNA assessment, the blood samples will be preserved appropriately. All AE(s) and SAE will be followed until resolution or the event is considered stable.

DETAILED DESCRIPTION:
The study is to compare treatment response of lamivudine and entecavir in patients with spontaneous severe acute exacerbation of chronic hepatitis B.

1. Primary objective:

• To compare the overall survival (OS) rate during observational period between lamivudine and entecavir therapy.

2. Secondary objectives:

1. To compare the change from baseline in HBV DNA level at each visit between lamivudine and entecavir therapy.
2. To compare the proportion of subjects who have a ≥ 2 log10 decline from baseline in HBV DNA level at each visit between lamivudine and entecavir therapy.
3. To compare the change from baseline in ALT and AST level at each visit between lamivudine and entecavir therapy.
4. To compare the proportion of subjects with prolonged prothrombin time (PT) at each visit between lamivudine and entecavir therapy.
5. To compare the change from baseline in bilirubin level at each visit between lamivudine and entecavir therapy.
6. To compare the transplantation-free survival rate during observational period between lamivudine and entecavir therapy.
7. To assess the safety of lamivudine and entecavir treatments in patients with HBV-associated severe acute exacerbation.

Statistical method(s) for safety/efficacy evaluations:

1. The major analysis will be performed according to the principal of intent-to-treat population; the safety evaluation will be performed according to the safety population.
2. For primary endpoint, the time to event will be analyzed by Kaplan-Meier method and summarized as the number of observations, number of censored, median time point estimate and the 95% CI for median.
3. Secondary efficacy endpoints:

1. Change from baseline in HBV DNA level at each visit 2. Proportion of subjects with HBV DNA response* at each visit

* Defined as a ≥ 2 log10 decline from baseline HBV DNA level. 3. Change from baseline in ALT level at each visit 4. Change from baseline in AST level at each visit 5. Proportion of subjects with prolonged PT* at each visit
* PT at each visit will also be assessed. 6. Change from baseline in bilirubin level at each visit 7. Transplantation-free survival rate during observational period Continuous variables will be analyzed using two-sample t-test/ Wilcoxon Rank Sum test, and categorical variables will be analyzed Chi-squared/ Fishers' exact test. Descriptive statistics including mean, standard deviation, median, minimum, maximum, 95% confidence interval will be also presented. Categorical variables will be summarized by counts and percentage in frequency table. In addition, the time to event will be analyzed by Kaplan-Meier method.

  (4) The summary results of laboratory at the baseline and the end of study visit, the change from baseline to end of study visit will be summarized by descriptive statistics and paired t-test will be used under significant level 0.05.

  (5) Adverse events will be coded with MedDRA and a summary frequency table of adverse events will be provided. The severity and relationship to study medication of adverse events will be summarized as well. Furthermore, if any serious adverse event had occurred, the brief summary about serious adverse event will be described and listed in tables.

  (6) All statistical tests will be two-side and evaluated at the 0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 20 years of age
2. HBsAg carrier with spontaneously severe acute exacerbation for whom the treatment with nucleoside and nucleotide reverse transcriptase inhibitor (NRTI) such as lamivudine and entecavir is medically recommended
3. Patients who fulfills all of the following criteria at screening:

   * documented HBsAg positive for at least 6 months or anti-HBc IgM negative
   * HBV DNA ≥ 2,000 IU/mL*

     * The blood sample will be collected at screening visit, but this criterion will be checked after obtaining lab result. For patients fulfill all other criteria, they can be enrolled immediately.
   * total bilirubin ≥ 2 mg/dL or prolonged prothrombin time (PT) ≥ 3 sec
   * serum ALT ≥ 10 x ULN
4. Patient with sufficient renal function defined as SCr ≤ 1.5 x ULN or ClCr ≥ 50 mL/min
5. Willing and able to sign a written informed consent

Exclusion Criteria:

1. Female who is pregnant/lactating
2. Patient with underlying liver cirrhosis classified as Child-Pugh class B or C
3. Patients with documented hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV) co-infection
4. Patients with uncontrolled malignancy
5. History or presence of alcohol or substance abuse within 1 year prior to the initiation of NRTI treatment
6. History of hypersensitivity to any ingredient of observational drugs (Zeffix® or Baraclude®)
7. Current use of medicine which may induce hepatotoxicity
8. Use of any antiviral therapy for HBV, such as interferon-α (IFN-α) and other nucleotide/nucleoside analogues, within 6 months prior to the initiation of NRTI treatment or exposure to any treatment for more than 3 months
9. Use of any chemotherapy or immunosuppressive agents within 12 months prior to the initiation of NRTI treatment
10. Use of any investigational product, including drug and invasive medical device, within 4 weeks prior to the initiation of NRTI treatment
11. Patient with any medical or psychiatric condition, including the presence of significant abnormal laboratory values, which is considered not suitable for this study by investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HBV DNA level at each visit | day 0、3、5、8±2、15±3、22±3、29±3、85±7、180±7
  To compare the change from baseline in HBV DNA level at each visit during observational period between lamivudine and entecavir therapy.

SECONDARY OUTCOMES:
Overall survival (OS) rate during observational period | Change from baseline (day0) to day 3、5、8±2、15±3、22±3、29±3、85±7、180±7
  To compare the overall survival (OS) rate between lamivudine and entecavir therapy.
Proportion of subjects with HBV DNA response at each visit | day 0、3、5、8±2、15±3、22±3、29±3、85±7、180±7
  To compare the proportion of subjects who have a ≥ 2 log10 decline from baseline in HBV DNA level at each visit between lamivudine and entecavir therapy.
Change from baseline in ALT and AST level at each visit | Change from baseline (day0) to day 3、5、8±2、15±3、22±3、29±3、85±7、180±7
  To compare the change from baseline in ALT and AST level at each visit between lamivudine and entecavir therapy.
Change from baseline in bilirubin level at each visit | Change from baseline (day0) to day 3、5、8±2、15±3、22±3、29±3、85±7、180±7
  To compare the change from baseline in bilirubin level at each visit between lamivudine and entecavir therapy.
Proportion of subjects with prolonged PT at each visit | day 0、3、5、8±2、15±3、22±3、29±3、85±7、180±7
  To compare the proportion of subjects with prolonged prothrombin time (PT) at each visit between lamivudine and entecavir therapy.
Transplantation-free survival rate during observational period | day 0、3、5、8±2、15±3、22±3、29±3、85±7、85±7、180±7
  To compare the transplantation-free survival rate during observational period between lamivudine and entecavir therapy.
To assess the safety of lamivudine and entecavir treatments in patients with HBV-associated severe acute exacerbation. | day 0 to day 180±7
  1. Change in laboratory data
  2. Adverse events
  3. Serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Shun Yang, M.D., Principal Investigator — Taichung Veterans General Hospital; Yu-Chun Hsu, M.D., Principal Investigator — Changhua Christian Hospital; Shih-Jer Hsu, M.D., Principal Investigator — National Taiwan University Hospital Yu-Lin Branch; Hsueh-Chou Lai, M.D., Principal Investigator — China Medical University Hospital; Chun-Che Lin, M.D., Principal Investigator — Chung Shan Medical University; Jen-Chieh Huang, M.D., Principal Investigator — ChengChing Hospital; Chi-Yi Chen, M.D., Principal Investigator — Chia-Yi Christian; Tsung-Ming Chen, M.D., Principal Investigator — Tung's Taiching MetroHarbor Hospital
Locations (8):
- Taiwan (8):
  - Changhua Christian Hospital, Changhua, Taiwan
  - Chia-Yi Christian, Chiayi City, Taiwan
  - Chung Shan Medical University Hospital, Taichung, Taiwan
  - China Medical University Hospital, Taichung, Taiwan
  - ChengChing Hospital, Taichung, Taiwan
  - Taichung Veterans General Hospital, Taichung, Taiwan
  - Tung's Taiching MetroHarbor Hospital, Taichung, Taiwan
  - National Taiwan University Hospital Yu-Lin Branch, YuLin, Taiwan

REFERENCES:
- [Derived] Lee TY, Chen CY, Lia HC, Hsu YC, Yang SS. The ultra-short virological dynamics in response to entecavir or lamivudine during chronic hepatitis B with spontaneous severe acute exacerbation. Antivir Ther. 2018;23(1):77-85. doi: 10.3851/IMP3183. PMID 28671553